CLINICAL TRIAL: NCT06321380
Title: Efficacy of Working Memory Maintenance Mechanisms in Alzheimer's Disease and Vascular Dementia
Brief Title: Working Memory Functioning in Alzheimer's Disease and Vascular Dementia
Acronym: MEMTRAV-COG
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Grenoble Alps (Other); Université Savoie Mont Blanc (Other); Centre National de la Recherche Scientifique, France (Other); Laboratoire de Psychologie et NeuroCognition (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC23.0381
Record Dates: First submitted 2024-02-05; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Alzheimer Disease; Vascular Dementia; Mixed Dementias
Keywords: Working memory; Alzheimer disease; Vascular dementia; Mixed dementia; Complex span task
MeSH Terms: conditions — Alzheimer Disease; Dementia, Vascular; Mixed Dementias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Alzheimer disease: Alzheimer's disease is define on the basis of the medical diagnostic. As part of routine care, they undergo a standardized clinical neuropsychological assessment that evaluates several cognitive functions.
  For the study and during the day of medical consultations, each patient will perform a working memory task, lasting approximately 30 minutes.
  If the patient is accompanied by a family member, the investigators ask the latter to complete a questionnaire on patient's daily executive functioning (French version of the Behavior rating inventory of executive function [BRIEF-A]).
  Interventions: Behavioral: Complex span task; Diagnostic Test: Clinical neuropsychological assessment
- Vascular dementia: Vascular dementia is define on the basis of the medical diagnostic. As part of routine care, they undergo a standardized clinical neuropsychological assessment that evaluates several cognitive functions.
  For the study and during the day of medical consultations, each patient will perform a working memory task, lasting approximately 30 minutes.
  If the patient is accompanied by a family member, the investigators ask the latter to complete a questionnaire on patient's daily executive functioning (French version of the Behavior rating inventory of executive function [BRIEF-A]).
  Interventions: Behavioral: Complex span task; Diagnostic Test: Clinical neuropsychological assessment
- Mixed dementia: Mixed dementia (i.e., Alzheimer's disease and vascular dementia) is define on the basis of the medical diagnostic. As part of routine care, they undergo a standardized clinical neuropsychological assessment that evaluates several cognitive functions .
  For the study and during the day of medical consultations, each patient will perform a working memory task, lasting approximately 30 minutes.
  If the patient is accompanied by a family member, the investigators ask the latter to complete a questionnaire on patient's daily executive functioning (French version of the Behavior rating inventory of executive function [BRIEF-A]).
  Interventions: Behavioral: Complex span task; Diagnostic Test: Clinical neuropsychological assessment
- Control group: Control group includes healthy older adults (without cognitive impairment). As patient group, control group will perform the working memory task. However, control group does not undergo the clinical neuropsychological assessment.
  Interventions: Behavioral: Complex span task; Diagnostic Test: Clinical neurospychological assessement

INTERVENTIONS:
Behavioral: Complex span task — The intervention consists in a computerized working memory task. This task follows the design of a complex span task, involving alternation between memorization and processing steps.
  For each trial, participants have to memorize French words. These words are sequentially displayed on the screen. Between each word, participants perform a processing task consisting in a spatial location task: They have to determine if a shape is at the top or at the bottom of the screen. After each processing episode, participants have a free time (i.e., available time to maintain information in WM). At the end of each trial, participants perform an orally immediate recall. This experimental task involves several conditions in order to manipulate the opportunities for the spontaneous use of refreshing and elaborative strategies.
  Other Names: Working memory task
Diagnostic Test: Clinical neuropsychological assessment — As part of routine care, participants in the patient group undergo a standardized clinical neuropsychological assessment that evaluates several cognitive functions. The investigators hypothesize correlations between working memory performance during the experimental task and the results of neuropsychological tests. Thus, the investigators consider the results to several French versions of neuropsychological tests:
  * MMSE (Mini-Mental State Examination)
  * "Digit Span Backward" subtest (WAIS-IV)
  * Stroop Test
  * Trail Making Test (TMT)
  * Rappel Libre - Rappel Indicé à 16 items or GERIA-12
  * Category fluences
  * Instrumental Activities of Daily Living and ADL .
  Groups: Alzheimer disease; Mixed dementia; Vascular dementia
Diagnostic Test: Clinical neurospychological assessement — Participants in the control group undergo 2 tests clinical that evaluate cognitive functioning.
  The investigators consider the results to French versions of these neuropsychological tests:
  * MMSE (Mini-Mental State Examination; )
  * "Digit Span Backward" subtest (WAIS-IV)
  Groups: Control group

SUMMARY:
The aim of the present study is to investigate potential cognitive mechanisms contributing to working memory impairment in Alzheimer's disease and vascular dementia. The investigators consider a new hypothesis suggesting that difficulties in mobilizing maintenance strategies of information could explain this working memory deficit. More specifically, the investigators assume that patient groups will have difficulties in employing both refreshing and elaborative strategies during a working memory task (i.e., complex span task), as compared to a control group.

DETAILED DESCRIPTION:
Working memory is considered as a central hub in human cognition. Good working memory capacities are fundamental for daily life. However, previous research has indicated that patients with Alzheimer's disease or vascular dementia have significant working memory impairment. Currently, there is no consensus on the cognitive mechanisms responsible for this deficit. Prior findings have highlighted that patients with Alzheimer's disease and/or vascular dementia demonstrate specific difficulties in dual-task situations. In this context, the investigators hypothesize that the continuous alternation between maintenance and processing phases involved in working memory could be impaired for these patients. Thus, the aim of the present study is to investigate if patients with Alzheimer's disease and/or vascular dementia can use maintenance strategies of information in working memory, as typically observed in individuals without cognitive impairments.

To this end, the investigators propose a short working memory task in which they manipulate the opportunities to use refreshing strategies and elaborative strategies. The investigators expect that patients with Alzheimer's disease, vascular dementia, or mixed dementia will benefit less than healthy older adults from the increased opportunities to employ refreshing and elaboration. These difficulties could account for the impaired working memory performance associated with these diseases.

In a second step, the investigators formulate distinctive hypotheses between patient sub-groups:

* On the one hand, Alzheimer's disease is characterized by salient impairment of episodic long-term memory. Consequently, the investigators hypothesize that the working memory decline could be related to this deficit in long-term memory. Specifically, patients with Alzheimer's disease would have greater difficulty in implementing elaboration strategies. Thus, these patients' recall performance should benefit less from semantic links between the to-be-remembered items compared to patients with vascular dementia.
* On the other hand, vascular dementia is characterized by a significant impairment of executive functioning. Thus, the investigators hypothesize that the working memory decline could be related to difficulties in implementing refreshing strategies (i.e., voluntary control of attention). Thus, the recall performance of these patients should benefit less from increased free time during the task, compared to patients with Alzheimer's disease.
* Finally, very few studies have been carried out on patients with mixed dementia (from both Alzheimer's disease and vascular dementia). The investigators assume that the recall performance of these patients will benefit less from elaborative opportunities compared to patients with dementia vascular, and less from refreshing opportunities compared to patients with Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* For patient and control groups: Adults ≥ 65 years of age
* For patient and control groups: Native French speaker
* For patient and control groups: Vision for easy reading
* For patient and control groups: Hearing for easy instruction understanding
* For patient and control groups: Back span ≥ 3 during the "Digit Span Backward" subtest (WAIS-IV)
* For patient and control groups: Formulation of the non-opposition to participate in this study
* For patient group only: Consultation in Grenoble University Hospital (Centre de Gérontologie Sud - Gerontology center) for clinical neuropsychological assessment due to suspected cognitive impairment
* For patient group only: Diagnosis of Alzheimer's disease, vascular dementia, or mixed dementia (i.e., Alzheimer's disease and vascular dementia)
* For patient group only: Have undergone a neuropsychological assessment at the day clinic, less than 6 months old.
* For patient group only: Have obtained a medical opinion stating that there is no contraindication to participate in this study and no concurrent pathology that could impair the patient's cognitive abilities.
* For patient group only: Absence of praxis and language disorders thath might prevent the carrying out of the experimental task.
* For patient group only: MMSE score between 18 and 25 included
* For control group only: External visitor/carer of a patient/resident of Grenoble University Hospital or volunteers at Grenoble University Hospital.
* For control group only: MMSE score ≥ 26

Exclusion Criteria:

* For patient and control groups: People under guardianship or deprived of their freedom
* For patient and control groups: Diagnosis of severe psychiatric disorders
* For patient and control groups: Suspicion of pathologies related to alcohol dependence
* For patient and control groups: No French social security coverage
* For patient and control groups: Refusal to voluntarily participate in this study
* For patient and control groups: People covered by articles L1121-5 to L1121-8 of the French Public Health Code
* For patient group only: Suspicion of another neurodegenerative disease, such as fronto-temporal dementia, Parkinson's disease, Lewy body disease.
* For patient group only: Clinical neuropsychological assessment did not reveal any cognitive impairment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The population of this study will consist of patients performing a neuropsychological assessment at Grenoble-Alpes University Hospital. These patients consult because of cognitive disorders. The patients are dividied into these three subgroups according to their medical diagnosis of Alzheimer's disease, vascular dementia, or mixed dementia (diagnostic criteria : Dubois et al. (2021) for Alzheimer's disease; VASCOG diagnostic criteria : Sachdev et al., 2015 for vascular dementia; and diagnostic criteria : DSM-V (APA, 2013) for mixed dementia due to Alzheimer and vascular etiology). The population of this study will also include healthy participants (carers/visitors of patients at the Gerontology centre or volunteers at Gerontology centre).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Memory performance in the Working memory task | 15 minutes
  Percentage of correct immediate recall, computed with strict serial recall criterion (item identity + correct position) and computed with item recall criterion (item identity only).
Processing performance in the Working memory task | 15 minutes
  Percentage of correct response in the spatial part of working memory task
Reaction time | 30 minutes
  Reaction time for each distractor (in ms) in the spatial part of working memory task

SECONDARY OUTCOMES:
Mini-Mental State Examination (MMSE) | 15 minutes
  MMSE is a test evaluate global cognitive functioning Score from 0 to 30 A higher score mean a better cognitive efficiency
Digit span forward WAIS IV (digit number) | 5 minutes
  The participant's span is noted, corresponding to the longest number of sequential digits that can be repeated forward.
Digit span forward WAIS IV (standard note) | 5 minutes
  This scale permitted to obtain a standard note from 0 to 19 A higher score means a better performance
Digit span backward WAIS IV (digit number) | 5 minutes
  The participant's span is noted, corresponding to the longest number of sequential digits that can be repeated backward.
Digit span backward WAIS IV (standard note) | 5 minutes
  This scale permitted to obtain a standard note from 0 to 19 A higher score means a better performance
Stroop Test - denomination part | 30 secondes
  the denomination part of stroop test measures processing speed time is taken, in seconds
Stroop Test - minor interference part (Time) | 30 secondes
  this part of stroop test measures low inhibition process time is taken, in seconds
Stroop Test - minor interference part (errors) | 30 secondes
  this part of stroop test measures low inhibition process number of errors is noted, from 0 to 24
Stroop Test - major interference part (time) | 90 secondes
  this part of stroop test measures strong inhibition process time is taken, in seconds
Stroop Test - major interference part (errors) | 90 secondes
  this part of stroop test measures strong inhibition process number of errors is noted, from 0 to 24
Trail Making Test - Part A (time) | 2 minutes
  This test evaluate motor speed processing Time in seconds
Trail Making Test - Part A (errors) | 2 minutes
  This test evaluates motor speed processing Number of errors is noted
Trail Making Test - Part B (time) | 5 minutes
  This test evaluates mental flexibility Time in seconds
Trail Making Test - Part B (errors) | 5 minutes
  This test evaluates mental flexibility Number of errors is noted
Category fluences | 5 minutes
  Number of correct words is noted
Memory evaluation (16-item Free and Cued Recall, or GERIA-12) | 40 minutes
  These tests evaluate verbal episodic memory Scores are noted for each trail, from 0 to 16 (RL-RI/16) or 0 to 12 (Geria-12) A higher score means a better performance
Naming task | 40 minutes
  This test evaluate the capacity to correctly name a picture Score is noted, from 0 to 40 A higher score means a better performance
Behavior rating inventory of executive function | 10 minutes
  Questionnaire (french version) on patient's daily executive functioning, completed by a relative of the patient, if present Global score from 75 to 225, composing by several composite scores. A higher score means a more severe executive dysfonctionning in daily life
Instrumental Activities of Daily Living | 5 minutes
  Questionnaire completed by a professional (nurse or doctor) with the patient and an accompagniant if present Score from 0 to 8 A higher score mean a better autonomy in daily life
Activities of Daily Living | 5 minutes
  Questionnaire completed by a professional (nurse or doctor) with the patient and an accompagniant if present Score from 0 to 6 A higher score mean a better autonomy in daily life

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Lemaire, Study Chair — Laboratoire de Psychologie et NeuroCognition; Sophie Portrat, Study Chair — Laboratoire de Psychologie et NeuroCognition

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartsch LM, Singmann H, Oberauer K. The effects of refreshing and elaboration on working memory performance, and their contributions to long-term memory formation. Mem Cognit. 2018 Jul;46(5):796-808. doi: 10.3758/s13421-018-0805-9. PMID 29557069
- [Background] Belleville S, Chertkow H, Gauthier S. Working memory and control of attention in persons with Alzheimer's disease and mild cognitive impairment. Neuropsychology. 2007 Jul;21(4):458-69. doi: 10.1037/0894-4105.21.4.458. PMID 17605579
- [Background] Camos V, Johnson M, Loaiza V, Portrat S, Souza A, Vergauwe E. What is attentional refreshing in working memory? Ann N Y Acad Sci. 2018 Jul;1424(1):19-32. doi: 10.1111/nyas.13616. Epub 2018 Mar 15. PMID 29542133
- [Background] Conway AR, Kane MJ, Bunting MF, Hambrick DZ, Wilhelm O, Engle RW. Working memory span tasks: A methodological review and user's guide. Psychon Bull Rev. 2005 Oct;12(5):769-86. doi: 10.3758/bf03196772. PMID 16523997
- [Background] Inasaridze K, Foley JA, Logie RH, Sala SD. Dual task impairments in vascular dementia. Behav Neurol. 2010;22(1-2):45-52. doi: 10.3233/BEN-2009-0252. PMID 20543458
- [Background] Zheng C, Zhang RS, Wan T, Zhao JS. Topological Alterations of Working Memory Impairment in Aged Patients With Vascular Dementia. Front Aging Neurosci. 2021 Oct 4;13:741445. doi: 10.3389/fnagi.2021.741445. eCollection 2021. PMID 34675799
- [Background] Baddeley AD, Baddeley HA, Bucks RS, Wilcock GK. Attentional control in Alzheimer's disease. Brain. 2001 Aug;124(Pt 8):1492-508. doi: 10.1093/brain/124.8.1492. PMID 11459742
- [Background] Belleville S, Peretz I, Malenfant D. Examination of the working memory components in normal aging and in dementia of the Alzheimer type. Neuropsychologia. 1996 Mar;34(3):195-207. doi: 10.1016/0028-3932(95)00097-6. PMID 8868277
- [Background] Foley JA, Cocchini G, Logie RH, Della Sala S. No dual-task practice effect in Alzheimer's disease. Memory. 2015;23(4):518-28. doi: 10.1080/09658211.2014.908922. Epub 2014 Apr 30. PMID 24787541
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Gagnon LG, Belleville S. Working memory in mild cognitive impairment and Alzheimer's disease: contribution of forgetting and predictive value of complex span tasks. Neuropsychology. 2011 Mar;25(2):226-36. doi: 10.1037/a0020919. PMID 21090897
- [Background] Jahn H. Memory loss in Alzheimer's disease. Dialogues Clin Neurosci. 2013 Dec;15(4):445-54. doi: 10.31887/DCNS.2013.15.4/hjahn. PMID 24459411
- [Background] Jellinger KA, Attems J. Prevalence and pathology of vascular dementia in the oldest-old. J Alzheimers Dis. 2010;21(4):1283-93. doi: 10.3233/jad-2010-100603. PMID 21504129
- [Background] KATZ S, FORD AB, MOSKOWITZ RW, JACKSON BA, JAFFE MW. STUDIES OF ILLNESS IN THE AGED. THE INDEX OF ADL: A STANDARDIZED MEASURE OF BIOLOGICAL AND PSYCHOSOCIAL FUNCTION. JAMA. 1963 Sep 21;185:914-9. doi: 10.1001/jama.1963.03060120024016. No abstract available. PMID 14044222
- [Background] Korczyn AD, Vakhapova V, Grinberg LT. Vascular dementia. J Neurol Sci. 2012 Nov 15;322(1-2):2-10. doi: 10.1016/j.jns.2012.03.027. Epub 2012 May 8. PMID 22575403
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] McGuinness B, Barrett SL, Craig D, Lawson J, Passmore AP. Executive functioning in Alzheimer's disease and vascular dementia. Int J Geriatr Psychiatry. 2010 Jun;25(6):562-8. doi: 10.1002/gps.2375. PMID 19810010
- [Background] O'Brien JT, Thomas A. Vascular dementia. Lancet. 2015 Oct 24;386(10004):1698-706. doi: 10.1016/S0140-6736(15)00463-8. PMID 26595643
- [Background] Raoux N, Le Goff M, Auriacombe S, Dartigues JF, Amieva H. [Semantic and letter fluency tasks: normative data in an elderly population of 70 years old and over from the PAQUID cohort]. Rev Neurol (Paris). 2010 Jun-Jul;166(6-7):594-605. doi: 10.1016/j.neurol.2010.01.012. Epub 2010 Mar 16. French. PMID 20236672
- [Background] Tombaugh TN. Trail Making Test A and B: normative data stratified by age and education. Arch Clin Neuropsychol. 2004 Mar;19(2):203-14. doi: 10.1016/S0887-6177(03)00039-8. PMID 15010086
- [Background] Vandenberghe M, Michiels J, Vanderaspoilden V, Claes T, Fery P. [Creation and normalisation of a verbal episodic memory task in elderly adults: "GERIA-12"]. Rev Neurol (Paris). 2015 Dec;171(12):853-65. doi: 10.1016/j.neurol.2015.08.001. Epub 2015 Nov 10. French. PMID 26563664
- [Background] Vergauwe E, Ricker TJ, Langerock N, Cowan N. What do people typically do between list items? The nature of attention-based mnemonic activities depends on task context. J Exp Psychol Learn Mem Cogn. 2019 May;45(5):779-794. doi: 10.1037/xlm0000625. Epub 2018 Jul 19. PMID 30024250
- [Background] Roy, A., Fournet, N., Le Gall, D., Roulin, J. L. BRIEF. Inventaire d'évaluation comportementale des fonctions exécutive - Adaptation française. Hogrèfe France Editions (2014).
- [Background] Logie, R., Camos, V., & Cowan, N. Working memory: State of the science. Oxford University Press. (2020).
- [Background] Grober E., & Buschke H. . Genuine memory deficits in dementia. Developmental Neuropsychology,(1987) 5, 13-36.
- [Background] Craik, F. I. M., & Tulving, E. Depth of processing and the retention of words in episodic memory. Journal of Experimental Psychology (1975). General, 104, 268-294.
- [Background] Bayard, S., Erkes, J., & Moroni, C. (2009). Test du Stroop Victoria-Adaptation Francophone. CPCN-LR, Gignac.